CLINICAL TRIAL: NCT04398264
Title: Characteristics of COVID-19 Infection Among PREGnant Women
Acronym: CCOVID-PREG
Status: Completed | Type: Observational
Sponsor: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Luis M. Gomez, Associate Professor, Inova Health Care Services
Other Study IDs: U20-05-4055
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Corona Virus Infection; Pregnancy Related
Keywords: COVID-19; SARS-Cov2; 2019-nCoV; Vertical transmission; Asymptomatic positive; Pandemics; Universal screening; Obstetric; Viral infection
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 positive via testing — Pregnant women admitted to Obstetric Units undergo RT-PCR testing for the detection of SARS-Cov2 (COVID-19 infection)

SUMMARY:
In December 2019, Coronavirus infection (COVID-19) was identified as causing serious respiratory infection in humans. Initially COVID-19 was propagated by infected symptomatic individuals; currently the disease is disseminated by asymptomatic COVID-19 positive subjects. The prevalence of asymptomatic COVID-19 individuals is unknown.

Due its physiologic immune suppression, pregnancy is a vulnerable time for severe respiratory infections including COVID-19.

Limited information is available regarding the impact of COVID-19 in pregnancy and the prevalence and demographic profile of asymptomatic pregnant women.

Despite reports of 15-20% positive COVID-19 tests in women admitted to Labor and Delivery, professional obstetric medical societies still recommend not prioritizing testing of patients who are asymptomatic.

In the USA, COVID-19 symptomatic patients come predominantly from lower income, Black and Latino communities. No data are available on the rate and demographic distribution of asymptomatic positive COVID-19 pregnant women.

To minimize the risk of inadvertent exposure asymptomatic individuals, recently our institution started COVID-19 testing in all admitted pregnant women. The investigators expect to gain knowledge on the impact of COVID-19 in pregnant women especially if asymptomatic and compare to other respiratory infections.

DETAILED DESCRIPTION:
TITLE: Characteristics of COVID-19 infection in pregnant women (CCOVID-PREG)

Background Coronavirus disease 2019 (COVID-19) is an infectious disease characterized by severe respiratory illness which can lead to multi-organ damage. It was reported in December 2019 in China, and was declared as a pandemic on March 11, 2020. The number of cases quickly increased in the USA since March; as of May 5th the total number of cases was 1'171,510 with 68,279 deaths.

COVID-19 is mainly spread through respiratory droplets of infected persons. While most respiratory viruses are more infectious when a patient is symptomatic, viral, epidemiology and modeling evidence suggest that also pre-symptomatic and asymptomatic individuals are able to transmit the infection. This information has implications on how resources can be spent on public interventions to prevent spreading of the virus. It also can help guide further management of pregnant women before, at, and after delivery.

Despite a recent publication reporting near 20% rate of positive COVID-19 tests in all pregnant women with a 13% rate of asymptomatic patients admitted to Labor and Delivery, the Society for Maternal Fetal Medicine and the Center for Disease Control and Prevention (CDC) still recommend not prioritizing testing of patients who are asymptomatic. Meanwhile, the American College of Obstetricians and Gynecologists published a recent Practice Advisory that encouraged prioritization of symptomatic patients but also acknowledges the potential impact of asymptomatic patients.

Racial disparities have been reported among non-pregnant adults infected with COVID-19. Lower income communities in New York City have a higher rate of infection, with Black and Hispanic communities found to be twice more likely to die from the infection as compared to Caucasians. Hispanic individuals are 1.7 more likely to get infected compared to their non-Hispanic peers. As many individuals in these communities are essential workers such as city employees and service personnel, many are undocumented; this is why public health interventions such as home isolation, social distancing, and early testing might not be applicable to these populations.

Inova Fairfax Hospital along with other hospitals from the Inova Health System (IHS) is located in the Washington District of Columbia (DC)-Northern Virginia-Maryland area in the east coast of the USA. Our hospitals provide obstetric care including anterpartum management, surgeries and delivery to a vast number of patients with private insurance as well as those uninsured from charity clinics in Northern Virginia. To minimize the risk of inadvertent exposure of non-infected pregnant women and health care personnel to COVID-19 positive asymptomatic patients, on April 25, 2020 IHS hospitals started testing for COVID-19 all pregnant women admitted to Labor and Delivery and Antepartum units. In our institution, the authors aim to investigate:

* Rate of COVID-19 positive pregnant women
* Prevalence of COVID-19 positive symptomatic and asymptomatic pregnant women admitted to obstetric services
* Demographic profile of COVID-19 positive asymptomatic pregnant women
* Clinical outcomes of COVID-19 positive symptomatic and asymptomatic women
* Rate of COVID-19 positive newborns from infected mothers
* Rate and profile of COVID-19 infected pregnant women who require respiratory support in comparison to those affected by other respiratory infections

Study design and participants This is an observational chart review study. Clinical records and compiled data of all hospitalized and outpatient pregnant women with laboratory-confirmed COVID-19 from March 18, 2020 to March 17, 2021 from IHS hospitals will be included in a database. COVID-19 is diagnosed on the basis of the CDC definition.[12] A confirmed case of COVID-19 is defined as a positive result on real-time reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay of nasal-pharyngeal swab specimens.[13] Data on recent exposure history, presence or absence of clinical symptoms or signs, laboratory findings, and maternal and perinatal outcomes will be collected. All medical records will be sent to the principal investigator at Inova Fairfax Hospital. Data will be entered into a computerized de-identified database and cross-checked.

Outcomes and Abstracted Data The main outcome of the study is the rate of asymptomatic pregnant women who test positive for COVID-19 at the time of hospital admission.

Secondary outcomes will be:

* Rate of Hispanic pregnant women among those asymptomatic COVID-19 positive on admission
* Rate of asymptomatic positive pregnant women who later will develop COVID-19 related symptoms
* Prevalence of COVID-19 positive newborns from infected mothers
* Rate of COVID-19 positive pregnant women who develop respiratory / multi-organ complications requiring admission to Medicine or Intensive Care units
* Rate of maternal death related to COVID-19 infection

Data to be obtained during chart abstraction will be:

Maternal:

* Demographics: Ethnicity, Age. Type of medical insurance, Preferred mode of transportation, Job information
* Body mass index
* Clinical indicators of mild disease: Fever, Cough, Abnormal sense of smell or taste, Shortness of Breath, Diarrhea
* Clinical indicators of moderate disease: Dyspnea, Pneumonia, Refractory Fever
* Clinical indicators of severe clinical course: Admission to intensive care unit (ICU), Acute Respiratory Distress Syndrome (ARDS), Need for mechanical ventilation, Multi-Organ Failure, Maternal Mortality
* Abnormal Laboratory Results: Leukopenia, Lymphopenia, Thrombocytopenia, Abnormal liver enzymes
* Obstetric outcomes: Spontaneous Abortion, Perinatal Mortality, Preterm delivery (PTD), Fetal growth restriction (FGR), Preeclampsia, Cesarean delivery (CD) Neonatal: Admission to neonatal intensive care unit (NICU), Rate of newborns testing positive for COVID-19 whose mothers are known COVID-19 infected individuals (symptomatic and asymptomatic), Vertical transmission, Apgar Scores, Breastfeeding

Statistical analysis The authors will use SAS 9.4 software (SAS Inc, Cary, NC) for our analyses. Data will be shown as means ± standard deviation (SD), or as medians (range), or as numbers (percentage).

ELIGIBILITY:
Inclusion Criteria:

* >18 years-old
* Pregnant women admitted to obstetric units (Labor and Delivery, Antepartum High Risk Pregnancy, pre-operative obstetric related surgeries as Cesarean or Cerclage) of Inova Health System hospitals

Exclusion Criteria:

- Pregnant women not tested for COVID-19

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Pregnant women who presented to our Institution during the study period
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Asymptomatic COVID-19 positive pregnant women | Through completion of the study, an average of 1 year
  Rate of asymptomatic pregnant women who test positive for COVID-19 at the time of hospital admission

SECONDARY OUTCOMES:
Asymptomatic Hispanic COVID-19 positive pregnant women | Through completion of the study, an average of 1 year
  Rate of Hispanic pregnant women among those asymptomatic COVID-19 positive on admission
Follow up of asymptomatic COVID-19 positive pregnant women | Through completion of the study, an average of 1 year
  Rate of asymptomatic positive pregnant women who later will develop COVID-19 related symptoms
COVID-19 positive newborns | Through completion of the study, an average of 1 year
  Prevalence of COVID-19 positive newborns from infected mothers
Severe COVID-19 disease in pregnant women | Through completion of the study, an average of 1 year
  Rate of COVID-19 positive pregnant women who develop respiratory / multi-organ complications requiring admission to Medicine or Intensive Care units / maternal death related to COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- INOVA Health System, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
Since COVID-19 in pregnant women is still a novel topic, we anticipate the need for collaboration with other researchers studying the effects of COVID-19 in pregnant women.
  Individual participant data that underlie the results to be reported in our research would be available to be shared after deidentification (text, tables, figures and appendices) for individual participant meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our Institution's data warehouse but without investigator support other than deposited metadata.
  Time Frame: Beginning 9 months and ending 36 months following article publication.
  Information to be shared: Study Protocol, Results.
  Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] CDC. Coronavirus Disease 2019 (COVID-19) in the U.S. Centers for Disease Control and Prevention. Published April 29, 2020. Accessed May 5, 2020. https://www.cdc.gov/coronavirus/2019-ncov/cases-updates/cases-in-us.html
- [Background] CDC. Coronavirus Disease 2019 (COVID-19) - Transmission. Centers for Disease Control and Prevention. Published April 13, 2020. Accessed May 5, 2020. https://www.cdc.gov/coronavirus/2019-ncov/prevent-getting-sick/how-covid-spreads.html
- [Background] Furukawa NW, Brooks JT, Sobel J. Evidence Supporting Transmission of Severe Acute Respiratory Syndrome Coronavirus 2 While Presymptomatic or Asymptomatic. Emerg Infect Dis. 2020 Jul;26(7):e201595. doi: 10.3201/eid2607.201595. Epub 2020 Jun 21. PMID 32364890
- [Background] Vintzileos WS, Muscat J, Hoffmann E, John NS, Vertichio R, Vintzileos AM, Vo D. Screening all pregnant women admitted to labor and delivery for the virus responsible for coronavirus disease 2019. Am J Obstet Gynecol. 2020 Aug;223(2):284-286. doi: 10.1016/j.ajog.2020.04.024. Epub 2020 Apr 26. No abstract available. PMID 32348743
- [Background] Vahidy FS, Nicolas JC, Meeks JR, Khan O, Pan A, Jones SL, Masud F, Sostman HD, Phillips R, Andrieni JD, Kash BA, Nasir K. Racial and ethnic disparities in SARS-CoV-2 pandemic: analysis of a COVID-19 observational registry for a diverse US metropolitan population. BMJ Open. 2020 Aug 11;10(8):e039849. doi: 10.1136/bmjopen-2020-039849. PMID 32784264